CLINICAL TRIAL: NCT06279377
Title: Evaluation of the Efficacy of Stabilization Exercise Training After Cervical Laminoplasty Surgery: A Randomized Controlled Study
Brief Title: Examining the Effectiveness of Exercise Training After Cervical Laminoplasty Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Sevtap Günay, Associate Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Katip Celebi University
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spine Disease; Surgery; Rehabilitation; Exercise
Keywords: Cervical Laminoplasty; Exercise Training; Stabilization Exercises; Early Exercise
MeSH Terms: conditions — Motor Activity | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization Exercise Group (Experimental): In the stabilization exercise group, in addition to those performed in the standard exercise group, training of deep neck flexor muscles with stabilizers and dynamic stabilization exercises will be applied.
  Stabilizer Pressure Biofeedback unite, elastic resistance bands and elastic balls will be used in the stabilization exercise program.
  Exercises performed with an elastic resistance band will be started in the 4th week, and exercises performed with an elastic ball will be started in the 6th week, depending on the suitability of the patient.
  Interventions: Other: Stabilization Exercises
- Standard Exercise Group (Active Comparator): On the day they will be discharged from the hospital, cervical normal joint movement, patient and posture training will be given.
  Then the exercise program will begin and the first session will be held. Patients will be given a 5-minute warm-up program before starting the exercise and a 5-minute cool-down program at the end of the exercise.
  Cervical flexion, extension, lateral flexion and rotation movements will be performed within the scope of the warm-up and cool-down program. Then, posture exercises and neck exercises with elastic resistance band will be performed.
  Interventions: Other: Standard Exercises

INTERVENTIONS:
Other: Stabilization Exercises — * Stabilizer Pressure Biofeedback device will be used in deep neck flexors training. Once the starting level is determined, training will be carried out with 2 mmHg pressure increases until the target value is 30 mmHg.
  * During the exercises performed with the elastic resistance band, the patient will be asked to move the band with his hands (neck extension, right-left lateral flexion).
  * During the exercises with the elastic ball, you will be asked to press your head on the ball at 90 degree angles (in 4 positions).
  * Exercises will be performed in 10 repetitions by maintaining muscle contraction for 10 seconds. Exercises will be performed as 1 set of 10 repetitions or 2 sets of 10 repetitions, depending on the patient's tolerance. When 2 sets are completed successfully, the color of the elastic resistance band or the level of the exercise will be changed and continued.
  Other Names: Experimental Group
  Arms: Stabilization Exercise Group
Other: Standard Exercises — * Cervical flexion, extension, lateral flexion and rotation movements will be performed within the scope of the warm-up and cool-down program. Cervical movements will be limited to approximately 30 degrees in the early period.
  * As posture exercises, you will be asked to do scapular retraction and turning your shoulders forward and backward. In addition to these movements, pectoral stretching, anterior and posterior capsule stretching exercises will be performed.
  * Elastic resistance bands will be used during neck exercises. Patients will be asked to perform cervical flexion, extension and right-left lateral flexion movements against the fixed band.
  * Patients will be asked to continue each exercise for 10 seconds. Exercises will be performed as 1 set of 10 repetitions or 2 sets of 10 repetitions, depending on the patient's tolerance. When 2 sets are completed successfully, the elastic resistance band color will be changed and the exercise will progress.
  Other Names: Active Comparator (Control) Group
  Arms: Standard Exercise Group

SUMMARY:
The goal of this clinical trial is to compare the effects of the stabilization exercise program applied after cervical laminoplasty surgery compared to standard exercise on pain, dysfunction, normal joint movement, proprioception, balance, muscle endurance, postural alignment and related factors (kinesiophobia, awareness, quality of life, disability, physical activity level). The main question[s] it aims to answer are:

* Does the exercise program applied after cervical laminoplasty surgery have an effect on pain, dysfunction, normal joint movement, proprioception, balance, muscle endurance, postural alignment and related factors (kinesiophobia, awareness, quality of life, disability, physical activity level)?
* Does the stabilization exercise program applied after cervical laminoplasty surgery have an effect on pain, dysfunction, normal joint movement, proprioception, balance, muscle endurance, postural alignment and related factors (kinesiophobia, awareness, quality of life, disability, physical activity level)?

Patients will start their first exercise session on the day they will be discharged from the hospital. Patients in both exercise groups will be provided with cervical normal joint movement (ROM), posture and patient education on the day of discharge. They will be asked to do posture exercises and neck exercises under the guidance of a physiotherapist. Patients in the stabilization exercise group (experiment) will undergo stabilization exercises under the supervision of a physiotherapist, in addition to the practices in the standard exercise group. Both groups will do a warm-up program before exercise and a cool-down program afterwards. Patients will be asked to do the exercises face to face with a physiotherapist 3 days a week. The first evaluations will be made on the day they come to the outpatient clinic for examination before surgery. Post-surgical evaluations will be made routinely after the exercise program is completed, when they are called by the physician for a check-up (6th week).

Researchers will compare the standard exercise group with the stabilization exercise group to see if pain, dysfunction, normal joint movement, proprioception, balance, muscular endurance, postural alignment and related factors (kinesiophobia, awareness, quality of life, disability, physical activity level) are different.

DETAILED DESCRIPTION:
Patients who are decided to undergo cervical laminoplasty surgery, whose eligibility is determined according to the inclusion and exclusion criteria, and who voluntarily agree to participate in the study will sign an informed consent form before the study begins. After consent is obtained, patients will be divided into 2 groups, standard exercise group and stabilization exercise group, by computer-assisted randomization method. As a result of the randomization, the evaluator will not know which group the patients belong to. Evaluations for all groups; It will be carried out twice, on the day they come to the polyclinic for pre-surgical examination, and on the 6th week after the surgery, when they are routinely called by the physician for a check-up.

In the first evaluation, sociodemographic information (age, gender, height, weight, BMI, occupation, curriculum vitae, family history), health-related habits (smoking, alcohol, exercise habits), dominant upper and lower extremity will be questioned. Pain intensity (VAS), dysfunction (mJOA score), normal joint movement (digital inclinometer), proprioception (Laser Assisted Angle Repetition Test), balance (Computerized balance platform), kinesiophobia (Tampa Kinesiophobia Questionnaire), level of awareness (Neck Awareness Questionnaire) quality of life (SF-12), disability (Neck Disability Index), physical activity level (IPAQ-short form) and radiographic findings regarding to postural alignment will be evaluated. Radiographic findings of the patients will be interpreted according to the results obtained from routine control evaluations before and after surgery.

Patients included in the standard exercise group; warming up and cooling down program, posture exercises and neck exercises will be applied for 6 weeks. For patients in the stabilization exercise group, in addition to the practices in the standard exercise group, deep neck flexors training with stabilizers and dynamic stabilization exercises with elastic resistance band and elastic ball will be performed. Training with stabilizer will be applied for 6 weeks. Elastic resistance band exercises will be performed in the 4th week, and exercises with an elastic ball will be applied starting from the 6th week until the end of the exercise program. The 'standard exercise group' constitutes the control group of the study and the 'stabilization exercise group' constitutes the experimental group. Patients in both groups will be given cervical normal joint movement, posture and patient education on the day they will be discharged from the hospital. The first exercise session will also be held on the day you are discharged from the hospital. Patients who are not seen on the day of discharge from the hospital will start an exercise program as soon as possible (within the first week following discharge).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cervical pathologies identified by clinical symptoms and imaging
* Patients who are indicated to undergo cervical laminoplasty by a specialist in spine surgery
* Volunteering to participate in the study
* Becoming literate in Turkish

Exclusion Criteria:

* Having had previous spine surgery
* Having any neurological, cardiopulmonary, orthopedic, metabolic, vestibular problems that may affect evaluation and exercise application
* Malignancy or spinal tumor
* Spine infection
* Fracture or traumatic subluxation of cervical vertebrae after surgical procedure
* Severe axial or extremity pain after surgery, presence of hyperesthesia that makes activity difficult, or extremity paralysis
* Not attending 3 consecutive exercise sessions or participating less than 80% in the total exercise session

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Preoperative and postoperative 6th week (at the end of the exercise program)
  Pain intensity will be assessed using the Visual Analogue Scale (VAS). While evaluating with VAS, patients will be asked to mark the degree of pain they feel on a 100 mm horizontal line.
Dysfunction | Preoperative and postoperative 6th week (at the end of the exercise program)
  It will be evaluated using the Modified Japanese Orthopedic Association (mJOA) Score, modified from the Japanese Orthopedic Association (JOA) score. It is a scale in which a total of 18 points can be obtained. Based on the mJOA score, 15-17 is defined as mild, 12-14 as moderate, and 0-11 as severe myelopathy. The recovery rate after surgery is calculated by the formula [Healing rate (%) = [(post-op JOA score - pre-op JOA score) / (18- pre-op JOA score)] X 100]. Recovery rate; >75% is considered excellent, 50-75% is considered good, 25-50% is inadequate, and <25% is considered poor.
Joint Range of Motion | Preoperative and postoperative 6th week (at the end of the exercise program)
  Active range of motion will be automatically calculated using the ACUMAR™ digital inclinometer. Cervical flexion, extension, right-left lateral flexion and right-left rotation movements of the patients will be evaluated.
Proprioception | Preoperative and postoperative 6th week (at the end of the exercise program)
  'Laser Assisted Angle Repetition Test', which is frequently used in the clinic, will be applied. The process will be repeated for cervical flexion, extension, right-left rotation and right-left lateral flexion. The error distance will be recorded and the tan value will be calculated.
Balance | Preoperative and postoperative 6th week (at the end of the exercise program)
  Balance assessment will be performed using a uniaxial force platform (ProKin 252, Tecnobody, Dalmine, Italy) with a sampling rate of 20 Hz and sensitivity of 0.1°. Static balance (eyes open and closed) and limit of stability will be evaluated.
Neck Extensor Muscle Endurance | Preoperative and postoperative 6th week (at the end of the exercise program)
  The digital inclinometer will be fixed to the lateral side of the head with velcro so that the screen of the device can be read. During the evaluation, patients will be asked to tuck their chin in and maintain the position by keeping their head in a horizontal alignment for as long as possible.
Neck Flexor Muscles Endurance | Preoperative and postoperative 6th week (at the end of the exercise program)
  During the test, the digital inclinometer will be fixed to the lateral side of the evaluator's head with velcro. Patients will be asked to lift their head approximately 2.5 cm (1 inch) off the bed by pulling their chin back and towards their chest (as if doing yes or no). Patients will be asked to maintain the position for as long as possible.
Postural Alignment | Preoperative and postoperative 6th week (at the end of the exercise program)
  Angular values obtained from routine radiographic findings of the patients will be calculated.

SECONDARY OUTCOMES:
Kinesiophobia | Preoperative and postoperative 6th week (at the end of the exercise program)
  It will be evaluated with the 'Tampa Kinesiophobia Scale'. The person receives a total score between 17-68. A high score on the scale indicates that the person's fear of movement is also high. The person receives a total score between 17 and 68. A high score on the scale indicates that the person has a high fear of movement.
Neck Awareness | Preoperative and postoperative 6th week (at the end of the exercise program)
  It will be evaluated with the Fremantle Neck Awareness Questionnaire. The total score of the survey is between 0-36. Higher scores indicate greater neck awareness.
Life Quality | Preoperative and postoperative 6th week (at the end of the exercise program)
  SF-12 Quality of Life scale will be used for evaluation. While the physical component summary (PCS)-12 score is obtained from the subscales of general health, physical functionality, physical role and body pain, the mental component summary (MCS)-12 score is obtained from the social functionality, emotional role, mental health and energy subscales. . Both the PCS-12 and MCS-12 scores range from 0 to 100, with a higher score representing better health.
Disability | Preoperative and postoperative 6th week (at the end of the exercise program)
  It will be evaluated with the Neck Disability Index. The patient's test score is determined according to certain score ranges: 0-4 (no disability), 5-14 (mild disability), 15-24 (moderate disability), 25-34 (severe disability), 35 and above (complete disability).
Physical Activity Level | Preoperative and postoperative 6th week (at the end of the exercise program)
  It will be evaluated using the International Physical Activity Questionnaire. Calculation of the total score includes the sum of the duration (minutes) and frequency (days) of walking, moderate activity and vigorous activity. There are three levels of physical activity identified when classifying populations categorically: 'inactive', 'minimally active' and 'very active' (physical activity that enhances health).

OTHER OUTCOMES:
Sociodemographic İnformation | Pre-surgery
  The sociodemographic information of the patients to be questioned includes age, gender, occupation, CV and family history.
Sociodemographic İnformation BMI | Pre-surgery
  The sociodemographic information of the patients to be questioned includes height, weight, BMI,
Health-related Habits | Pre-surgery
  Health-related habits to be questioned include smoking and alcohol use, exercise habits.
Dominant Side | Pre-surgery
  It will be obtained by questioning the patients' dominant use of their lower and upper extremities during specific activities.

CONTACTS AND LOCATIONS:
Overall Officials: Sevtap GUNAY UCURUM, Assoc. Dr., Study Director — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University Ataturk Education and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No